CLINICAL TRIAL: NCT01763749
Title: Comparison of the Efficacy and Safety of Closone and Clopidogrel With Aspirin in Korean Patients With Coronary Artery Disease (a Single-center, Randomized, Open-label Clinical Trial)
Brief Title: Comparison of the Efficacy and Safety of Closone and Clopidogrel With Aspirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Kiyuk Chang, Associate professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLO_1201
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closone (Experimental): 75mg/100mg per day, 4weeks, PO
  Interventions: Drug: Closone
- Plavix with Astrix (Active Comparator): Plavix 75mg with Astrix 100mg, 4weeks, PO
  Interventions: Drug: Plavix with Astrix

INTERVENTIONS:
Drug: Closone — Closone 75mg/100mg, 4weeks, PO
  Arms: Closone
Drug: Plavix with Astrix — Plavix 75mg with Astrix 100mg, 4weeks, PO
  Arms: Plavix with Astrix

SUMMARY:
The Aim of this study is to prove non-inferiority of Closone to the Combination treatment of Plavix with Astrix.

ELIGIBILITY:
Inclusion Criteria:

* Subjects under condition after Post-Percutaneous Coronary Artery Intervention over twelve months
* 20~85 years old
* Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

* Subject who did not undergo or failed Stent Implantation
* Subjects who took an anti-coagulant, anti-thrombotic regularly before the study, or plan to have continuous treatment during the study
* Subjects with a history of hypersensitivity to Clopidogrel, Aspirin
* Subjects with uncontrolled severe hypertension
* Subjects with high risk of hemorrhage like blood coagulation disorders

  :gastrointestinal bleeding, gross hematuria, intraocular bleeding, hemorrhagic stroke, intracranial hemorrhage
* Subjects with intractable arrhythmia, intracranial hemorrhage
* Subjects with Severe cardiomyopathy (New York Heart Association(NYHA) Class Ⅳ)
* Subjects with Severe hepatopathy(AST and ALT > 10 times the upper limit of normal)
* Subjects who are pregnant, breastfeeding and not using medically acceptable birth control
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in P2Y12% inhibition at week 4 | Baseline, week 4

SECONDARY OUTCOMES:
Change from baseline in VerifyNow P2Y12 reaction unit at week 4 | Baseline, week 4
  PRU : VerifyNow P2Y12 reaction unit
Change from baseline in VerifyNow Aspirin Reaction Unit at week 4 | Baseline, week 4
  ARU : VerifyNow Aspirin Reaction Unit
Change from baseline in maxymal platelet aggregation at week 4 | Baseline, week 4
  MPA : maxymal platelet aggregation

OTHER OUTCOMES:
Adverse events | Baseline, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, MD, PhD, Principal Investigator — Cardiovascular center and Cardiology Division, Seoul St. Mary's Hospital
Locations (1):
- Cardiovascular Center and Cardiology Division, Seoul St. Mary's Hospital, Seoul, Seochogu, South Korea